CLINICAL TRIAL: NCT01787838
Title: A Quality Improvement Study to Improve Pneumococcal Vaccination Rates Through Targeted Health Education for Patients in an Ambulatory Pre-surgical Testing Setting
Brief Title: Improving Pneumococcal Vaccination Rates in an Ambulatory Pre-surgical Testing Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carilion Clinic (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Clark_Merck_2.4.2013
Record Dates: First submitted 2013-02-04; First posted 2013-02-11 (Estimated); Results first posted 2014-08-26 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Community Acquired Pneumonia
Keywords: Pneumococcal vaccination rates, ambulatory settings
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- health education, audit and feedback (Other): Focused health education for staff and patients.
  Interventions: Other: Focused Health Education

INTERVENTIONS:
Other: Focused Health Education — A two-phase quality improvement study was designed to modify staff and patient behaviors. The project incorporated evidence-based strategies of staff education, feedback and incentives for performance and patient education.
  The staff received monthly feedback on departmental immunization rates, and incentives for performance. A one-page patient education flyer, written at 3rd grade reading level, was added to encourage patients to inquire about it.
  Other Names: Patient literature and staff education, reinforcement

SUMMARY:
The purpose of this quality improvement project is to improve the immunization rates of an at-risk adult population seen in an ambulatory healthcare environment, through the use of targeted health education messages regarding pneumococcal immunization. Patients seen in an out-patient pre-surgical testing center will receive 1) a one-page written information sheet that outlines the benefits of pneumococcal immunization and 2) verbal reinforcement of this message, provided by the clinical staff, during the patient's interview.

At-risk adult patients (as defined by Centers for Disease Control) seen in an ambulatory healthcare environment (a pre-surgical testing center) will receive a one page, "gain-framed" message that emphasizes the benefits of pneumococcal vaccinations. This educational material will be reviewed and reinforced by clinical staff during the assessment phase of the clinical visit. Among this group, there will be increased vaccination rate compared with at-risk adult patients who did not receive this communication (prospective vs retrospective data).

DETAILED DESCRIPTION:
The purpose of this project was to improve the immunization rates of an at-risk adult population seen in an ambulatory environment, through the use of targeted and evidence-based health education messages regarding pneumococcal immunization and staff training on the use of gain-framed messaging.

We hypothesized that there would be an increase in immunization rates for at-risk adults following implementation of the intervention.

The objective of the project was to increase our local immunization rate by 30% (from 20% to 50%) and to provide tools and processes that can be utilized in other ambulatory healthcare settings.

ELIGIBILITY:
Inclusion Criteria:

* Patient seen in out-patient pre-surgical testing center
* At-risk adult patient as defined by the Centers for Disease Control (CDC)

Exclusion Criteria:

* Minors

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2509 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca C Clark, PhD, Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Clinic, Roanoke, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients seen in the presurgical testing center who were eligible were offered the pneumococcal vaccine.
Groups:
- Health Education, Audit and Feedback: Prospective single group intervention with retrospective control group with no intervention.
  Focused Health Education: A two-phase quality improvement study was designed to modify staff and patient behaviors. The project incorporated evidence-based strategies of staff education, feedback and incentives for performance and patient education.
  The staff received monthly feedback on departmental immunization rates, and incentives for performance. A one-page patient education flyer, written at 3rd grade reading level, was added to encourage patients to inquire about it.
Period: Overall Study
Arm/Group | Health Education, Audit and Feedback
Started | 2509 (This is the number who met Centers for Disease Control and Prevention guidelines for vaccine.)
Completed | 1096 (This is the number of patients successfully immunized in a one year period.)
Not Completed | 1413
Not completed — refused | 1413

BASELINE CHARACTERISTICS:
Population: All patients greater than 18 years of age, chronic diseases, smoker seen in presurgical testing center
Arm/Group | Health Education, Audit and Feedback
Number analyzed (Participants) | 2509
Age, Continuous [Mean (Full Range); unit: years] | 57 [19 to 84]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1757
  >=65 years | 752
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1531
  Male | 978
Region of Enrollment [Number; unit: participants]
  United States | 2509

OUTCOME MEASURES:

1. Primary Outcome: Improving Pneumococcal Vaccination Rates Following Focused Health Education of Staff and Patients
Description: Pneumococcal vaccination rates, tracked biweekly, following 1) staff education, audit and feedback of rates and 2) patient education
Time Frame: 12 Months
Measure: Number; unit: participants
Groups:
- Health Education, Audit and Feedback: Prospective single group intervention Focused Health Education: A two-phase quality improvement study was designed to modify staff and patient behaviors. The project incorporated evidence-based strategies of staff education, feedback and incentives for performance and patient education.
  The staff received monthly feedback on departmental immunization rates, and incentives for performance. A one-page patient education flyer, written at 3rd grade reading level, was added to encourage patients to inquire about immunizations.
Arm/Group | Health Education, Audit and Feedback
Number analyzed (Participants) | 2509
participants | 1096 [1.65 to 1.96]
Statistical Analysis 1: Comparison: Health Education, Audit and Feedback; Prospective data from 12 months were compared to data that had been collected for the previous 12 month period to determine statistical significance and trended outcomes for comparative periods. Patients were screened for eligibility during the first 12 months, and staff and patients received the interventions during the second 12 month period; Test type: Superiority or Other; p < .0001, Chi-squared; Odds Ratio (OR) = 1.80, 95% CI 2-sided [1.65 to 1.96]

ADVERSE EVENTS:
Time Frame: Time of visit to presurgical center
Arm/Group | Health Education, Audit and Feedback
Serious Adverse Events (participants affected / at risk) | 0/2509
Other Adverse Events (participants affected / at risk) | 0/2509

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No